CLINICAL TRIAL: NCT00744003
Title: Early Trauma Induced Coagulopathy (ETIC): A Pilot Study to Determine Its Definition and Risk Factors
Brief Title: An Observational Study of Early Coagulopathy, or Clotting Disorder, in Injured Patients
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer at Emory; no participants enrolled, study not conducted
Sponsor: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006685; ETIC Study (Other: Other)
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Trauma-induced Coagulopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Trauma continues to be the major killer of young Americans, mainly due to hemorrhage or brain injury. In trauma centers, up to a quarter of these severely injured patients arrive with a coagulopathy and thereby experience an increased risk of death, despite the current standard of medical and surgical management. The PI for this grant proposal is a fellowship-trained trauma surgeon who works full-time at Grady Memorial Hospital (GMH), the only Level I Trauma Center in Atlanta. It is only one of four Level 1 trauma centers for the entire state of Georgia. This research is a direct extension of the retrospective research the PI has previously published. Her retrospective research discovered a previously undescribed form of coagulopathy, early trauma induced coagulopathy (ETIC), which cannot be explained by present paradigms. Two civilian trauma articles as well as military data from the Iraq war have substantiated the occurrence of ETIC, but no prospective literature has defined it or its kinetics. More importantly, the results from these studies represent a new paradigm shift, in which ETIC appears to be a primary dysfunction which is independently associated with death. Therefore, its early identification and correction is crucial for our mechanistic understanding, and ultimately, our choice of interventions and improved survival. GMH is a high-volume trauma center that sees patients with a variety of injury mechanisms, and, therefore, is the perfect setting to confirm ETIC. First, the project will confirm the prevalence of ETIC with an observational prospective cohort of injured patients. Data on the coagulation system and risk factors, both known and suspected, of all patients will be collected upon patient arrival as well as patient outcome with all identifying information protected. This is the first prospective research project that will allow simultaneous control of confounders associated with outcome and thereby scientifically validate the occurrence of ETIC. One unique component of our data collection is a focus on the timing of events as they relate to the development and consequences of coagulopathy, to account for the dynamic process. At the completion of data collection, a matched cohort of ETIC and non-ETIC blood samples will be tested for coagulation factors to provide insight into ETIC's pathophysiology. In the short term, our conclusions will assist us in our approach to resuscitation of the bleeding trauma patient as some trauma centers have already started to change protocols based on our present incomplete understanding of trauma-induced coagulopathy. In addition, the coagulation system data collected in this study will lead to pathophysiological answers and to more refined hypotheses for future research at a coagulation system level. Ultimately an understanding of ETIC will lead to a more effective, tailored treatment. Our main study hypothesis is that post-trauma coagulopathy is a primary dysfunction that occurs early after a traumatic event in up to 25% of all trauma patients triaged to Trauma Center care.

ELIGIBILITY:
Inclusion Criteria:

1. > 17 years of age
2. GMH Emergency Care Center (ECC) admission with trauma team activation - referred to by GMH nomenclature as a "STAT-pack." Trauma team activation criteria were developed from standard criteria published by the American College of Surgeons Committee on Trauma and published in Resources for Optimal Care of the Injured Patient manual 2006 edition and modified for GMH use. A trauma patient is declared a STAT-pack if they meet one of the following criteria:

   * Ejection from a motor vehicle or motorcycle
   * Extremes of age: pediatric < 6 years of age or an adult > 65 yrs of age
   * One of the following: HR > 120; RR > 30; Systolic BP < 100; GCS < 13; Basal temperature < 35 degrees C
   * Penetrating trauma to head/neck/thorax/abdomen including flank and back/antecubital fossa/groins/popliteal space
   * Suspected neurological injury i.e. spinal cord injury
   * Traumatic amputation above the wrist or ankle
   * Mangled or crush to an extremity
   * History of trauma in a patient who is combative, has deteriorating vital signs or is hemorrhaging from an open wound
   * Physician or EMS discretion
3. Patients admitted to GMH ECC directly from the site of injury

Exclusion Criteria:

1. < 18 years of age
2. Any patient who is pronounced dead by health care personnel prior to any blood sampling
3. Any patient who arrives undergoing CPR and is pronounced dead without resumption of vital signs
4. Transfers from other health care facilities
5. Any patient known to be taking anti-coagulant or anti-platelet medicine
6. Any patient with a known predisposing history of a coagulation or platelet defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients arriving at a Level I trauma center who activated the Trauma Team criteria for a "stat pack" trauma admission
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Development of coagulopathy as defined by abnormal PT/INR | Admission to Trauma Center

CONTACTS AND LOCATIONS:
Overall Officials: Jana BA MacLeod, MD, Principal Investigator — Assistant Professor Of Surgery, Emory University School of Medicine
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States